CLINICAL TRIAL: NCT06035627
Title: Uncontrolled Inadvertent Perioperative Hypothermia as a Risk Factor for Surgical Site Infection in Patients Undergoing Laparoscopic Cholecystectomy: A Randomized Controlled Trial
Brief Title: The Effect of Inadvertent Perioperative Hypothermia on Surgical Site Infection in Laparoscopic Choleistectomy.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cumhuriyet University (Other)
Responsible Party: Principal Investigator, Pınar YILMAZ EKER, Asst. Prof, Cumhuriyet University
Other Study IDs: PYILMAZEKER
Record Dates: First submitted 2023-08-28; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Surgical Site Infection; Perioperative Complication
Keywords: inadvertent perioperative hypothermia; surgical site infection; laparoscopic cholecystectomies; perioperative nursing
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental group: The population of the study consisted of patients who were being treated in the general surgery clinic of the hospital, who met the sampling criteria, who were to undergo laparoscopic cholecystectomy, and who agreed to participate in the study. The sample size of the study was determined by the G*Power 3.1.9.7 program. In the power analysis, when α =0.05, β=0.10, and 1-β =0.90, the sample size was determined as 50 people per group and a total of 100 people.
  Interventions: Other: Prevention hypothermia
- Control group: The population of the study consisted of patients who were being treated in the general surgery clinic of the hospital, who met the sampling criteria, who were to undergo laparoscopic cholecystectomy, and who agreed to participate in the study. The sample size of the study was determined by the G*Power 3.1.9.7 program. In the power analysis, when α =0.05, β=0.10, and 1-β =0.90, the sample size was determined as 50 people per group and a total of 100 people.

INTERVENTIONS:
Other: Prevention hypothermia — Hypothermia was prevented by warming the case group. control group remained stable. As a result, the presence of surgical site infection was followed.
  Groups: Experimental group

SUMMARY:
There are conflicting results in the literature explaining the relationship between surgical site infection (SSI) and inadvertent perioperative hypothermia (IPH). Although it is thought that the risk of IPH is lower in laparoscopic surgery types due to the short duration of the surgical procedure, these conflicting results raise doubts as to whether there is a relationship between IPH and SSI in laparoscopic surgery patients. A randomized controlled study will be planned in the future to examine the effect of IPH on SSI in patients who will undergo laparoscopic cholecystectomies. The study will be conducted in the general surgery clinic and operating room of a university hospital. It will be completed with a total of 100 patients, 50 of whom will be in the case group, and 50 will be in the control group.

DETAILED DESCRIPTION:
Objective: This study was conducted to examine the effect of inadvertent perioperative hypothermia (IPH) on Surgical Site Infection (SSI) in patients undergoing laparoscopic cholecystectomy.

Summary of Background Data: There are conflicting results in the literature explaining the relationship between SSI and IPH. Although the risk of IPH is thought to be lower in laparoscopic surgery types due to the short duration of the surgical procedure, these conflicting results raise doubts about the existence of a relationship between IPH and SSI in laparoscopic surgery patients.

Methods: This study will be a quasi-experimental and randomized controlled study in the future. The study will be conducted with patients who will have undergone laparoscopic cholecystectomy in the general surgery clinic and operating room of a university hospital. The study will be completed with a total of 100 patients, 50 in the case group, and 50 in the control group. During the study, preoperative, intraoperative, and postoperative body temperatures, as well as biomarkers of the patients, will be monitored using a form developed by the researchers. Additionally, patients will be followed up postoperatively to evaluate the potential impact of IPH on SSI.

ELIGIBILITY:
Inclusion Criteria:

* Being aged 18-65 years old,
* Having an ASA score of I-II,
* Remaining in the hospital for at least 24 hours in the postoperative period,
* Undergoing laparoscopic cholecystectomy

Exclusion Criteria:

* Being under 18 or over 65,
* Having an ASA score above III,
* Requiring emergency surgery
* Having a neurological, psychiatric, or neuromuscular disease,
* Being addicted to alcohol and/or other toxic substances,
* Being pregnant or having a suspected pregnancy,
* Undergoing open surgery, or being converted to an open procedure during surgery,
* Having symptoms of fever
* Having an active infection excluding cholecystitis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: laparoscopic cholecystectomy patients who met the inclusion and exclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-15 (Actual); Primary Completion 2024-05-15 (Estimated); Study Completion 2024-08-15 (Estimated)

PRIMARY OUTCOMES:
Prevention of inadvertent perioperative hypothermia | September 15, 2022- September 15, 2023
  This study aims to evaluate whether inadvertent perioperative hypothermia has an effect on surgical site infection. For this, applications to prevent hypothermia will be applied to the patients in the experimental group

SECONDARY OUTCOMES:
Following surgical site infection | 16 September 16, 2023 - October 25, 2023
  After the applications for preventing hypothermia in the experimental group and the patients in the experimental and control groups will be examined for surgical site infection.

CONTACTS AND LOCATIONS:
Overall Officials: Pınar YILMAZ EKER, Ph.D, Principal Investigator — corresponding researcher
Locations (2):
- Turkey (Türkiye) (2):
  - Cumhuriyet University, Sivas, Suşehri
  - Sivas Cumhuriyet University, Sivas

REFERENCES:
- [Background] Connelly L, Cramer E, DeMott Q, Piperno J, Coyne B, Winfield C, Swanberg M. The Optimal Time and Method for Surgical Prewarming: A Comprehensive Review of the Literature. J Perianesth Nurs. 2017 Jun;32(3):199-209. doi: 10.1016/j.jopan.2015.11.010. Epub 2016 Sep 1. PMID 28527547
- [Background] Horn EP, Bein B, Broch O, Iden T, Bohm R, Latz SK, Hocker J. Warming before and after epidural block before general anaesthesia for major abdominal surgery prevents perioperative hypothermia: A randomised controlled trial. Eur J Anaesthesiol. 2016 May;33(5):334-40. doi: 10.1097/EJA.0000000000000369. PMID 26555870
- [Background] Scott AV, Stonemetz JL, Wasey JO, Johnson DJ, Rivers RJ, Koch CG, Frank SM. Compliance with Surgical Care Improvement Project for Body Temperature Management (SCIP Inf-10) Is Associated with Improved Clinical Outcomes. Anesthesiology. 2015 Jul;123(1):116-25. doi: 10.1097/ALN.0000000000000681. PMID 25909970
- [Background] Sessler DI. Perioperative thermoregulation and heat balance. Lancet. 2016 Jun 25;387(10038):2655-2664. doi: 10.1016/S0140-6736(15)00981-2. Epub 2016 Jan 8. PMID 26775126
- [Background] Ryczek E, White J, Poole RL, Reeves NL, Torkington J, Carolan-Rees G. Normothermic Insufflation to Prevent Perioperative Hypothermia and Improve Quality of Recovery in Elective Colectomy Patients: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2019 Dec 20;8(12):e14533. doi: 10.2196/14533. PMID 31859685
- [Background] Chen HY, Su LJ, Wu HZ, Zou H, Yang R, Zhu YX. Risk factors for inadvertent intraoperative hypothermia in patients undergoing laparoscopic surgery: A prospective cohort study. PLoS One. 2021 Sep 23;16(9):e0257816. doi: 10.1371/journal.pone.0257816. eCollection 2021. PMID 34555101